CLINICAL TRIAL: NCT01184794
Title: Postoperative Pain Control Using Continuous Infusion of Levobupivacaine in Women Undergoing Pelvic Operative Laparoscopy: A Randomised Controlled Trial
Brief Title: Postoperative Pain Control Using ON-Q Painbuster Pump
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ashford and St. Peter's Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008JTW01
Record Dates: First submitted 2010-06-18; First posted 2010-08-19 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Post Operative Analgesia
Keywords: Analgesia laparoscopy
MeSH Terms: interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline (Placebo Comparator): Placebo solution
  Interventions: Drug: levobupivacaine
- levobupivacaine, analgesia (Experimental): Active drug
  Interventions: Drug: levobupivacaine

INTERVENTIONS:
Drug: levobupivacaine — 40 ml over 48 hours
  Other Names: Chirocaine

SUMMARY:
This study is a blinded randomised study of slow release levobupivacaine vs saline for women undergoing day case operative pelvic laparoscopy. Participants will be randomly given either saline or levobupivacaine and efficacy will be measured using ranked ordinal pain scales and rescue oral analgesia use.

DETAILED DESCRIPTION:
METHOD:

This is a triple-blinded randomised control study to determine whether a continuous intraperitoneal infusion of levobupivacaine 0.5%, when compared with normal saline 0.9%, in women undergoing laparoscopic pelvic surgery as day-case, provides effective postoperative analgesia.

Primary outcome measure:

• Need for 'rescue' analgesia

Secondary outcome measures:

* Pain intensity (on movement and rest)
* Side effects from rescue analgesia
* Hospital length of stay
* Patient satisfaction with pain relief

Sample:

All women undergoing pelvic laparoscopic surgery as a day-case will be invited to take part in the study. Women will be excluded if they are undergoing surgery for cancer.

At the pre-operative admission clinic women will receive written information explaining the trial and inviting them to take part. If they agree to take part, written consent will be obtained on the morning that they arrive in the day ward for the laparoscopic procedure. At the end of the intended laparoscopic procedure, the peritoneal cavity will be irrigated with normal saline and then all the irrigation fluid will be removed through suction. The multihole catheter will then be inserted percutaneously into the surgical area although it will not be fixed into place. The catheter will be guided into place with the grasper or irrigator so that the holed portion of the catheter is in the intended area for anaesthetic infusion. The catheter will then be kept in place using a steri-strip to skin. Finally, the laparoscopic trocar sites will be closed in the usual way. Women will be randomised to receive either normal saline 0.9% or levobupivicaine 0.5%. Patients will be randomised at the start of the procedure so that the infusion can be prepared in time to be started at the end of the procedure. Randomisation will be undertaken using computer-generated random numbers, which will be held off site. The syringes and reservoir bladders Page 2 of 5 Version no. - 2 12.10.08

will be consecutively numbered and randomly filled with either levobupivacaine or normal saline using block randomisation in blocks of 10 to ensure equal number in each group. This will ensure that the surgeons, the anaesthetist and the patient will be blinded to the treatment group. In the event of an untoward incident the code will be broken, a sealed list being kept on the labour ward cupboard where it will be available 24 hours a day . At the end of the surgical procedure, a bolus of 5mls of the infusion will be delivered via the catheter, following which the rate is set at 2ml per hour. Patients will be discharged home in the usual way but will continue with the infusion for a total of 48 hours. Appropriate training will be in place for the participants and a leaflet will be given to them for support which will provide them with written instructions about the infusion device, how to care for it and how to remove it after the 48 hour period. They will also be provided with a telephone contact in case of any concerns about the infusion. Women who do not feel confident in removing the catheter at home will be requested to attend the gynaecology ward to have it removed by the gynaecology senior house officer. The participants will be provided with emergency contact telephone numbers if there are any concerns.

Power Calculation:

The sample size has been calculated based on the results of the randomised controlled study of bupivicaine versus normal saline in women undergoing an abdominal hysterectomy (Gupta et al 2004). In Gupta's study, the bupivicaine group used a total of 30.5mg (SD 15.4) of ketobemidone in the first 24 hours postoperatively. This compares to the placebo group, who used 44.3mg (SD 21.6); a clinically significant difference of approximately 30% reduction in pain in the treatment group.

Assuming an alpha of 0.05, we require a total of 52 patients (26 in each arm) to achieve a power of 90% (Beta = 0.1).

Page 3 of 5 Version no. - 2 12.10.08

Data collection:

All information relating to postoperative pain will be collected in a specifically designed pain measurement booklet. This will be completed whilst in hospital and then taken home with the patient for completion in the remaining 48 hours following surgery. The pages relating to pain measures experienced in hospital will be recorded on duplicate paper so that one copy can be retained in the medical records. Patients will be provided with a stamped addressed envelope for returning the pain measurement booklet.

Data to be collected:

All analgesia used will be recorded by amount and time taken. Pain will be measured at rest and on movement (walking and coughing) using a 10-point scale and will be taken at 1, 2, 3 and 4 hours. Thereafter the participants will be requested to record the pain intensity on the evening of the operation, morning-after the operation, afternoon on the following day, evening on the following day and on the second day after the operation i.e. 48 hours postoperatively. Time 0 will be taken to represent the time the infusion was started. Nausea will be measured on a 10-point scale and will be taken at for the 48 hour period while recording the pain intensity. Hospital length of stay will be recorded in hours and charted on the pain measurement booklet. Patient satisfaction will also be recorded as less than satisfied; satisfied; good or excellent. All patients will be contacted by telephone 48 hours postoperatively to enquire about their experiences of using the infusion device and to request them to return the pain measurement booklet.

Data Analysis:

Significance will be at the p=0.05 or less. SPSS software will be used to undertake the analysis under the supervision of Mr. Robert Hills.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing 'Day case' operative laparoscopic procedures.
* These women are deemed suitable to return home on the day of surgery, both in terms of physical fitness and their home circumstances.

Exclusion Criteria:

* Women having laparoscopic procedures for diagnostic purposes or minor operations such as sterilisation, will be excluded from the study.
* These procedures are less likely to cause significant pain due to operation.

Ages: 16 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Rescue analgesia use | 48 hours
  participants will record number of doses of oral analgesic tablets they required.

SECONDARY OUTCOMES:
Pain intensity on movement and rest | 48 hours
  participants are asked to complete a 10 point ranked ordinal pain score

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy T Wright, MD, Principal Investigator — Ashford and St. Peter's Hospitals NHS Trust
Locations (1):
- Ashford & St Peter's Hospitals NHS Trust, Chertsey, Surrey, United Kingdom